CLINICAL TRIAL: NCT06288893
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of SHEN211 Tablets in the Treatment of Patients With Mild and Moderate Novel Coronavirus Infection
Brief Title: SHEN211 Tablets for the Treatment of Mild and Moderate Novel Corona Virus Infections (COVID-19)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: JKT Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEU-2001
Record Dates: First submitted 2024-02-29; First posted 2024-03-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: SHEN211 tablets; multicenter phase II clinical study; efficacy; safety and pharmacokinetics
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized 2:1 to experimental and placebo arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHEN211 Tablets (Active Comparator): A total of 20 subjects were randomized to the test group
  Interventions: Drug: SHEN211 Tablets
- Placebo for SHEN211 Tablets (Placebo Comparator): 10 subjects randomized to placebo
  Interventions: Procedure: Placebo for SHEN211 Tablets

INTERVENTIONS:
Drug: SHEN211 Tablets — SHEN211 tablets, participants will receive 330 mg (3 tablets) QD (once a day) on Day 1 and 110 mg (1 tablet) SHEN211 tablets QD orally on Days 2-5.
  Other Names: Test group
  Arms: SHEN211 Tablets
Procedure: Placebo for SHEN211 Tablets — Placebo tablets, participants will receive 3 tablets QD (once daily) on Day 1 and 1 tablet QD orally on Days 2-5
  Other Names: control group
  Arms: Placebo for SHEN211 Tablets

SUMMARY:
Randomized, double-blind, placebo-controlled, multicenter phase II clinical study of SHEN211 tablets

DETAILED DESCRIPTION:
A total of 30 patients with mild to moderate novel coronavirus infection (COVID-19) were enrolled and randomized in a 2:1 ratio to the experimental and placebo groups, and subjects received 5 days of oral administration of SHEN211 or SHEN211 placebo to assess the effectiveness of SHEN211 tablets in the treatment of mild to moderate COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. subjects must be 18 years of age or older at the time of signing the informed consent form;
2. subject has a positive SARS-CoV-2 test result;
3. Subjects have one or more mild and moderate COVID-19 clinical symptoms with a symptom score of ≥ 2 (see Attached Table 2): fever, cough, sore throat or dry throat, nasal congestion or runny nose, fatigue or fatigue, headache, muscle or body pain (or soreness), shortness of breath or dyspnea, nausea, vomiting, diarrhea; Presence of one or more of the following signs/symptoms within 24 hours prior to randomization: fever, cough, sore throat or dry throat, nasal congestion or runny nose, fatigue or fatigue, headache, muscle or body aches (or aches), shortness of breath or dyspnea, nausea, vomiting, diarrhea;
4. subjects need to meet conditions: 1) The first occurrence of COVID-19 symptoms ≤ 3 days from the first administration of investigational product; 2) Samples for the first positive SARS-CoV-2 virus infection assay were ≤ 5 days from the first administration of investigational product; 3) SARS-CoV-2 viral nucleic acid detection Ct value ≤ 30 on the day of the first dose;
5. Subjects (women and men of childbearing age) and their sexual partners are willing to have no fertility plan and voluntarily take effective contraceptive measures and have no sperm donation or egg donation plan from the signing of the informed consent form to 1 month after the last dose of the study drug (see Appendix 6 for the definition and contraceptive measures of women of childbearing age);
6. The subject is able to understand and abide by the procedures and methods of this clinical trial. After full informed consent, the subject voluntarily participates and signs the informed consent form by himself/herself, or has a legal representative who can provide the informed consent form.

Exclusion Criteria:

1. subjects may progress to severe and severe COVID-19 before randomization as judged by the investigator;
2. SpO2 ≤ 93% or PaO2/FiO2 ≤ 300 mmHg, or respiratory rate ≥ 30/minute on sea-level room air;
3. urgent or expected need for nasal high-flow oxygen therapy or noninvasive positive pressure ventilation, invasive mechanical ventilation, or ECMO;
4. known history of active hepatitis (acute or chronic active hepatitis B or C), cirrhosis, or hepatic decompensation (including ascites, variceal bleeding, or hepatic encephalopathy); impaired immune system (including patients who have been treated with immunosuppressive agents for a long time, or patients with progressive or recurrent cancer, or known human immunodeficiency virus infection);
5. Screening ALT or AST > 1.5 times ULN or Cockcroft-Gault defined known current renal impairment as CrCl < 30 mL/min or requiring dialysis (see Appendix 4 for calculation formula);
6. Subjects who have received antiviral drugs (e.g., neltamivir tablets/ritonavir tablets, azvudine tablets, monoprevir capsules, sinotervir tablets/ritonavir tablets, deuterated remidavir hydrobromide tablets, and Chinese herbal medicine/Chinese patent medicine for anti-coronavirus therapy) treatment or prevention within 30 days before randomization;
7. The subject has received SARS-CoV-2 monoclonal antibody therapy or prophylaxis or antiviral therapy (including study treatment) or the subject has received convalescent COVID-19 plasma therapy;
8. the subject has a history of dysphagia or gastrointestinal disease that seriously affects drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, subtotal gastrectomy, etc.);
9. acute attack of chronic respiratory diseases, including bronchial asthma, chronic obstructive pulmonary disease;
10. concurrent influenza at screening, which may interfere with the assessment of response to study intervention based on symptoms, signs, laboratory tests, or imaging indicating a high likelihood of bacterial infection;
11. received any COVID-19 vaccine within 3 months before randomization, or infected with novel coronavirus within 3 months before randomization;
12. Complications requiring surgery before randomization or throughout the study period and major surgery 14 days before randomization, or life-threatening complications within 30 days before randomization as considered by the investigator;
13. Use of the following drugs within 14 days before enrollment: strong cytochrome P453A (CYP3A) inhibitors, strong CYP3A inducers, products containing St. John 's wort (Hypericum perforatum);
14. Participated in other clinical trials or taking experimental drugs within 3 months before randomization;
15. known hypersensitivity to any component used in the formulation of the intervention drug;
16. Pregnant and lactating women;
17. Patients who are judged by the investigator to be inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SARS-CoV-2 viral load at each time point | Up to day 28
  Change from baseline in SARS-CoV-2 viral load at each time point

SECONDARY OUTCOMES:
Time of recovery | Up to day 28
  To assess the time to first sustained recovery of 5/7/11 clinical symptoms (defined as time from first dose to COVID-19 symptom score of 0 and two days) in mild and moderate COVID-19 patients
Time to response | Up to day 28
  To assess time to first sustained resolution of 5/7/11 clinical symptoms (defined as time from first dose to COVID-19 symptom score of 0 or 1 and lasting 2 days) in mild and moderate COVID-19 patients
Time to negative | Up to day 28
  Time to Positive Viral Nucleic Acid Test to Negative
Percentage of subjects with disappearance of clinical symptoms | Up to day 28
  Percentage of subjects with disappearance of clinical symptoms on Days 1, 3, 5, 7, 10, 14, 21, and 28
Change in COVID-19 symptom score | Up to day 28
  Change in COVID-19 symptom score from baseline to Days 1, 3, 5, 7, 10, 14, 21, and 28
Ct value change from baseline | Up to day 28
  Change from baseline in SARS-CoV-2 Ct values on Days 1, 3, 5, 7, 10, 14, 21 and 28
Change from baseline in chest CT scan (optional) | Up to day 28
  Change from Baseline in Chest CT Scan on Days 3, 7, or 10 (Optional)
Percentage of Subjects Progressed | Up to day 28
  Percentage of subjects with COVID-19 progression (progression defined as severe/critical COVID-19 or death due to any cause) by Day 28
Percent of Subjects Who Died | Up to day 28
  Percentage of subjects with all-cause mortality by Day 28
Safety Assessment Results | Up to day 28
  Safety assessments (eg, AEs and SAEs) through Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, ph.D, Principal Investigator — Shenzhen Third People 's Hospital; Rui Song, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Shenzhen Third People 's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No